CLINICAL TRIAL: NCT04092595
Title: A PHASE 1, 2-PERIOD FIXED SEQUENCE, MULTIPLE-DOSE, OPEN-LABEL STUDY TO ESTIMATE THE EFFECT OF PF-06651600 ON ROSUVASTATIN PHARMACOKINETICS IN HEALTHY PARTICIPANTS
Brief Title: A Study of PF-06651600 Effect on Rosuvastatin Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7981024; 2019-002536-85 (EudraCT Number)
Record Dates: First submitted 2019-09-12; First posted 2019-09-17 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics (PK)
MeSH Terms: interventions — PF-06651600; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06651600 and Rosuvastatin (Experimental): Period 1 is 4 days in length. On Day 1 of Period 1 participants will receive a single dose of Rosuvastatin 10 mg given as a tablet orally. Period 2 is 11 days in length and will immediately follow Period 1 with no washout. In Period 2, participants will be dosed with oral 200 mg PF-06651600 once-daily (QD) for 7 days. On Day 8 of Period 2, a single dose of 10 mg Rosuvastatin oral tablet will be administered following administration of the 200-mg dose of PF-06651600. Dosing with oral 200 mg PF-06651600 QD will continue until Day 10 of Period 2.
  Interventions: Drug: PF-06651600; Drug: Rosuvastatin

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600: 200 mg dose provided as four 50 mg oral tablets
Drug: Rosuvastatin — 10 mg oral tablet
  Other Names: Crestor ®

SUMMARY:
A phase 1, 2-period, fixed-sequence, multiple-dose, open-label study of the effect of PF-06651600 on Rosuvastatin pharmacokinetics in healthy participants. Approximately 12 healthy male and/or female participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants who are healthy as determined by medical evaluation including medical history, full physical examination which includes blood pressure (BP) and pulse rate measurement, clinical laboratory tests, and 12-lead ECG.
* Body mass index (BMI) of 17.5 to 30.5 kg/m sq, and a total body weight greater than 50 kg (110 lb.).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Participants with any of the following acute or chronic infections or infection history:
* Any infection requiring treatment within 2 weeks prior to the dosing visit.
* Any infection requiring hospitalization, parenteral antimicrobial therapy within 60 days of the first dose of rosuvastatin.
* Any infection judged to be an opportunistic infection or clinically significant by the investigator, within the past 6 months of the first dose of rosuvastatin.
* Known active or history of recurrent bacterial, viral, fungal, mycobacterial or other infections.
* History of recurrent (more than one episode of) localized dermatomal herpes zoster, or history of disseminated (single episode) herpes simplex or disseminated herpes zoster.
* Known presence or a history of malignancy other than a successfully treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for rosuvastatin | Period 1 (4 days) day 1 and period 2 (11 days) day 8 , 0 (pre-dose), 0.5, 1,2,3,4,5,6,8,10,12,16,24,36,48,and 72 hours post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Renal clearance (CLr) for rosuvastatin | Period 1 (4 days) day 1 and period 2 (11 days) day 8 , hours: [0-6], [6-12], [12-24], [24-48], and [48-72] post-dose
  CLr = total amount of drug collected in urine (Ae) divided by area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981024